CLINICAL TRIAL: NCT04353427
Title: Improving Physical, Mental, and Spiritual Health in Faith-Based Settings Through Creating a Healthy Culture in Bronx, NY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-01617
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Mental Health Issue
MeSH Terms: interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Faith based educational group (Experimental): A seven-session faith-based small group educational program using the "The Seven Pathways to Healing, Health and Wellness" curriculum will be delivered.
  Interventions: Behavioral: The Seven Pathways to Healing, Health and Wellness curriculum

INTERVENTIONS:
Behavioral: The Seven Pathways to Healing, Health and Wellness curriculum — The curriculum seeks to increase civic engagement by fostering a sense of community and a sense of social and personal responsibility in community. There will be 7 monthly session that will be approximately 1 hour in duration. Session topics include:
  1. Education and Information (including mental health awareness, and a one-day certificate program in Mental Health First Aid)
  2. Connection with Others
  3. The Body as Temple
  4. Emotional Healing
  5. The Nature of Mind
  6. Life Assessment
  7. The Nature of Spirit

SUMMARY:
The proposed study "Improving Physical, Mental, and Spiritual Health in Faith- Based Settings through Creating a Healthy Culture in Bronx, NY" aims to assess the efficacy of a holistic health intervention that seeks to integrate physical, mental, spiritual, and community engagement processes into faith-based settings, compared to usual care in Bronx, NY. Briefly, the intervention involves a seven-session faith-based small group education program conducted by trained lay educators. A health ministry at each partner religious institution will be developed and sustained

DETAILED DESCRIPTION:
The purpose of this research study is test a holistic health intervention that combines physical, mental, spiritual, and community processes into faith-based settings in Bronx, NY. The program involves a seven-session faith-based small group education sessions to be conducted by lay educators.

ELIGIBILITY:
Intervention study participants

Inclusion Criteria:

* Age 18 and over
* Self-identify as a member of the religious institution for at least three months
* Able to read and speak in English, Vietnamese, or Khmer

Exclusion Criteria:

* Any serious health issue that may interfere with the study procedures

Key informants participants

Inclusion Criteria:

* Age 18 and over
* Must be a study implementation partner, a health ministry member, or lay educator

Exclusion Criteria:

* None

Focus group participants

Inclusion Criteria:

* Must be a participant in the intervention
* Attended at least 3 out of the 7 group education sessions as an intervention participant;

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in sociodemographic characteristics of participants | baseline and 6 months visit
  This will be measured by self reported participant survey about the aspects of personal and social responsibility for well-being.

SECONDARY OUTCOMES:
Facilitators and Barriers in intervention process by Focus Group participants | 6 months
  A Focus group of a subset of participants will assess the facilitators and barriers in receiving the 7 sessions of the intervention. The focus groups at a private location convenient for participants. Interviews will not exceed two hours and will be audio-recorded. The focus group data will elicit facilitators and barriers to receiving the intervention and making change to improve well-being. The focus group will discuss topics such as how the group sessions impacted on the participants' physical or mental health, what was challenging or not useful and what types of tools were gained that were helpful to become more spiritually healthy.
Facilitators and Barriers in intervention process by Key informants | 6 months
  The key informant interviews will contain questions that assess facilitators and barriers to implementing the intervention. The key informant interviews will be conducted once, immediately after completion of the intervention among intervention participants

CONTACTS AND LOCATIONS:
Overall Officials: Sahnah Lim, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request, Requests should be directed to Sahnah.lim@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.